CLINICAL TRIAL: NCT06117774
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Tarlatamab Therapy in Subjects With Limited-Stage Small-Cell Lung Cancer (LS-SCLC) Who Have Not Progressed Following Concurrent Chemoradiation Therapy
Brief Title: Study Evaluating Tarlatamab After Chemoradiotherapy in Limited-Stage Small-Cell Lung Cancer (LS-SCLC)
Acronym: DeLLphi-306
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230016; 2023-506235-15 (Other: EU CT Number)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Limited Stage Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: Limited Stage Small Cell Lung Cancer; Small Cell Lung Cancer; LS SCLC; SCLC; AMG 757; Tarlatamab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AMG 757

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tarlatamab (Experimental): Participants will receive tarlatamab on Cycle 1 Day 1, 8 and 15, and once every 2 weeks (Q2W) thereafter (cycle is 28 days).
  Interventions: Drug: Tarlatamab
- Placebo (Placebo Comparator): Participants will receive placebo on Cycle 1 Day 1, 8 and 15, and Q2W thereafter (cycle is 28 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tarlatamab — Intravenous (IV) infusion
  Other Names: AMG 757
  Arms: Tarlatamab
Drug: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the efficacy of tarlatamab with placebo as assessed by progression free survival (PFS) based on blinded independent central review (BCIR) per response evaluation criteria in solid tumors v1.1 (RECIST 1.1) and on prolonging overall survival (OS).

ELIGIBILITY:
Inclusion Criteria: -Participants are eligible to be included in the study only if all of the following criteria apply:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years).
* Histologically or cytologically confirmed small-cell lung cancer (SCLC).
* Diagnosed and treated for LS-SCLC with concurrent chemotherapy and radiotherapy.
* Has completed chemoradiotherapy without progression per RECIST 1.1 (ie, achieved complete response [CR], partial response [PR], or stable disease [SD]).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Minimum life expectancy of 12 weeks.
* Adequate organ function.
* Toxicities attributed to concurrent chemoradiotherapy resolved to grade ≤ 1, unless otherwise specified. Excluding alopecia or fatigue.

Exclusion Criteria: -Participants are excluded from the study if any of the following criteria apply:

Disease Related

* Extensive-stage SCLC (ES-SCLC).
* Any previous diagnosis of transformed non-small-cell lung cancer (NSCLC), epidermal growth factor receptor (EGFR) activating mutation positive NSCLC that has transformed to SCLC, or mixed SCLC NSCLC histology.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis. Other Medical Conditions
* History of other malignancy within the past 2 years, with certain exceptions.
* History of solid organ transplantation.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 6 months prior to first dose of study treatment.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 6 months prior to first dose of study treatment.
* Exclusion of human immunodeficiency virus (HIV) or active hepatitis infection based on criteria per protocol.
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.

Prior/Concomitant Therapy

* Received sequential chemotherapy and thoracic radiotherapy (no overlap of thoracic radiotherapy with chemotherapy) during chemoradiation.
* Prior therapy with any selective inhibitor of the delta-like ligand 3 (DLL3) pathway.
* Prior history of severe or life-threatening events from any immune-mediated therapy.
* Receiving another anti-cancer therapy. Adjuvant hormonal therapy for resected breast cancer is permitted.
* Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* Major surgical procedures within 28 days prior to first dose of study treatment.
* Treatment with live virus, including live-attenuated vaccination, within 14 days prior to the first dose of study treatment. Inactive vaccines and live viral non-replicating vaccines within 3 days prior to first dose of study treatment.

Prior/Concurrent Clinical Study Experience

• Treatment in an alternative investigational trial within 28 days prior to enrollment.

Other Exclusions

* Female participants of childbearing potential unwilling to use protocol specified method of contraception during treatment and for an additional 60 days after the last dose of study treatment.
* Female participants who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of study treatment.
* Female participants planning to become pregnant or donate eggs while on study through 60 days after the last dose of study treatment.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose of study treatment.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of study treatment.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of study treatment.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2030-05-29 (Estimated); Study Completion 2030-05-29 (Estimated)

PRIMARY OUTCOMES:
PFS as Determined by BICR | Up to approximately 6 years
OS Over the Whole Trial | Up to approximately 6 years

SECONDARY OUTCOMES:
PFS Determined by Investigator Assessment | Up to approximately 6 years
Objective Response (OR) Rate | Up to approximately 6 years
Disease Control (DC) Rate | Up to approximately 6 years
Duration of Response (DOR) | Up to approximately 6 years
PFS at 6 months, 1 year, 2 years | 6 months, 1 year, 2 years
OS at 6 months, 1 year, 2 years, 3 years | 6 months, 1 year, 2 years, 3 years
Time to Progression (TTP) | Up to approximately 6 years
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 6 years
Serum Concentration of Tarlatamab | Up to approximately 4 months
Incidence of Anti-tarlatamab Antibody Formation | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (203):
- United States (18):
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Los Angeles, Santa Monica, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Boca Raton Clinical Research Global South Florida, Plantation, Florida
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Our Lady of the Lake Cancer Institute, Baton Rouge, Louisiana
  - Morristown Medical Center, Morristown, New Jersey
  - New York University Grossman School of Medicine and New York University Langone Hospitals, New York, New York
  - Perlmutter Cancer Center at New York University Langone Hospital - Long Island, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Spokenword Clinical Trials, Easton, Pennsylvania
  - Renovatio Clinical, The Woodlands, Texas
  - US Oncology Research Investigational Products Center, The Woodlands, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - West Virginia University Health Sciences Center, Morgantown, West Virginia
- Argentina (8):
  - Fundacion Respirar, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Instituto Oncologico de Cordoba Ionc Fundacion Richardet Longo, Córdoba, Córdoba Province
  - Hospital Aleman Buenos Aires, CABA, Distrito Federal
  - Clinica Viedma, Viedma, Río Negro Province
  - Sanatorio 9 de Julio Cice 9 de Julio, San Miguel de Tucumán, Tucumán Province
  - Instituto Argentino de Diagnóstico y Tratamiento, Buenos Aires
- Australia (5):
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Brazil (15):
  - Hospital Santa Rita, Vitória, Espírito Santo
  - Oncoclinicas Onco Vida Distrito Federal, Brasília, Federal District
  - Liga Paranaense do Combate ao Cancer - Hospital Erasto Gaertner, Curitba, Paraná
  - Londrina Cancer Hospital, Londrina, Paraná
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Cipo - Centro Integrado de Pesquisa em Oncologia, Porto Alegre, Rio Grande do Sul
  - Centro de pesquisa em oncologia Hospital Ana Nery, Santa Cruz do Sul, Rio Grande do Sul
  - Centro Catarinense de Pesquisa LTDA, Blumenau, Santa Catarina
  - Fundacao pio xII Barretos, Barretos, São Paulo
  - Fundacao Amaral Carvalho, Jaú, São Paulo
  - Cepho, Santo André, São Paulo
  - Instituto Dor de Pesquisa e Ensino, Rio de Janeiro
  - Instituto Cancer Sao Paulo Icesp, São Paulo
- Bulgaria (7):
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagyurishte
  - Complex Oncology Center Plovdiv EOOD, Plovdiv
  - Complex Oncology Center Shumen EOOD, Shumen
  - University Multiprofile Hospital for Active Treatment Sofiamed OOD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- China (23):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Northern Jiangsu Peoples hospital, Yangzhou, Jiangsu
  - Jiangxi Cancer hospital, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Zhejiang Taizhou Hospital, Taizhou, Zhejiang
- Colombia (5):
  - Centro de Tratamiento e Investigación sobre Cancer Luis Carlos Sarmiento Angulo Ctic, Bogota, Cundinamarca
  - Instituto Nacional de Cancerologia, Bogota, Cundinamarca
  - Instituto Medico de Alta Tecnologia sas - Imat sas, Montería, Departamento de Córdoba
  - Oncologos del Occidente SAS, Pereira, Risaralda Department
  - Fundacion cardiovascular de Colombia, Bucaramanga, Santander Department
- France (5):
  - Centre Hospitalier Régional Universitaire de Lille - Institut Coeur Poumon, Lille
  - Centre Hospitalier Universitaire Nord, Marseille
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Nord Ouest Villefranche sur Saone, Villefranche-sur-Saône
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsmedizin Goettingen, Göttingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (7):
  - Agios Savvas Anticancer Hospital, Athens
  - Henry Dunant Hospital Center, Athens
  - Sotiria General Hospital, Athens
  - Attikon University Hospital, Athens
  - Metropolitan Hospital, Athens
  - Saint Luke Hospital, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Italy (10):
  - Centro di Riferimento Oncologico di Aviano, Aviano PN
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Istituto Oncologico Europeo, Milan
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Unita Sanitaria Locale di Reggio Emilia Arcispedale Santa Maria Nuova, Reggio Emilia
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Ospedale San Giuseppe Moscati, Statte
- Japan (20):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-Shi, Saitama
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Mexico (4):
  - Centro Oncologico Personalizado, Cuauhtémoc, Mexico City
  - Oncare, Mexico City, Mexico City
  - Oncocenter Clinica Integral Internacional de Oncologia, Puebla City
  - Phylasis Clinicas Research Toluca, Toluca
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Centrum Pulmonologii i Torakochirurgii w Bystrej, Bystra
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii imienia Eugenii i Janusza Zeylandow, Poznan
  - Szpital Specjalistyczny w Prabutach Spolka z Ograniczoną Odpowiedzialnoscia, Prabuty
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
- Portugal (3):
  - Unidade Local de Saude de Braga, EPE, Braga
  - Hospital da Luz, SA, Lisbon
  - Hospital Cuf porto, Porto
- Romania (7):
  - Spitalul Clinic de Urgenta Prof Dr Agrippa Ionescu, Balotesti, Ilfov
  - Institutul Oncologic, Prof Dr Alexandru Trestioreanu, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - SC Oncomed SRL, Timișoara
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Icon - Mount Alvernia, Singapore
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju Chungbuk
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Cha Bundang Medical Center, Cha University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (15):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Institut Catala d Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Instituto Valenciano de Oncologia, Valencia, Valencia
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Norrlands Universitetssjukhus, Umeå
- Switzerland (3):
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - Ospedale Regionale di Bellinzona e Vali, Mendrisio
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (12):
  - Ankara Etlik Sehir Hastanesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Dr Suat Seren Gogus Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Medical Park Seyhan Hastanesi, Mersin
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (2):
  - Guys Hospital, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com